CLINICAL TRIAL: NCT06865053
Title: Screening for Heart Failure in General Medicine Consultations (FIL-EAS ic Depistage)
Brief Title: Screening for Heart Failure in General Medicine Consultations
Acronym: DEPISTAGE IC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Cerballiance (Unknown); Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-003
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
Keywords: heart failure; screening; general medicine; care pathway; Multi-professional cooperation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients participating in the heart failure screening pathway in general medicine consultations
  Interventions: Other: Heart failure screening pathway

INTERVENTIONS:
Other: Heart failure screening pathway — Heart failure screening pathway in general medicine consultations (questionnaire, NT-proBNP level, echocardiographic examination)

SUMMARY:
Heart failure poses a significant public health challenge due to its high prevalence and the substantial human and financial costs it generates. Furthermore, the lack of clear screening guidelines and challenges in accessing care and multi-professional coordination, contribute to diagnostic delays, leading more patients to seek care in more severe clinical states and requiring direct admission to emergency departments. There is therefore also a major organizational challenge in better managing the entry of patients into the healthcare system. This necessitates the development of structured heart failure screening strategies.

The 2021 European Society of Cardiology (ESC 2021) guidelines on heart failure screening prioritize the identification of at-risk individuals and the early detection of disease manifestations. They suggest that, in high-risk groups, tests such as echocardiography and biomarker measurement (NT-proBNP) should be used to detect heart failure at an early stage, even in the absence of symptoms. The guidelines also delineate specific biomarker thresholds and propose organizational frameworks with defined timelines to facilitate systematic screening.

The implementation of a heart failure screening pathway within primary care involving multi-professional cooperation is therefore warranted.

Stratifying screening based on risk factors and symptomatology is expected to enhance the positive predictive value of the screening process. Furthermore, evaluating the efficacy of this pathway is crucial for establishing a standardized, reproducible clinical protocol suitable for routine primary care practice.

This study is a prospective, multicenter, observational study conducted within the context of routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consulting in general practice.
2. Aged 65 years or older

Exclusion Criteria:

1. Known heart failure.
2. Patient who has already consulted a cardiologist within the last 12 months.
3. Patient opposition to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years or older participating in the heart failure screening pathway in general medicine consultations
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of patients with a confirmed diagnosis of heart failure | 2 months
  i.e. patients with at least one "yes" box checked in "step 1" and "step 2" of the questionnaire, with an NT-proBNP level ≥ 125 pg/ml, and an echocardiographic examination performed by the cardiologist confirming a diagnosis of HF according to the 2021 ESC guidelines.
Rate of patients with an unconfirmed diagnosis of heart failure | 2 months
  i.e. all of the following patients:
  * Patients with no "yes" boxes checked in steps 1 and 2 of the questionnaire OR one or more "yes" boxes checked but in only one of steps 1 or 2.
  * Patients with at least one "yes" box checked in "step 1" and "step 2" of the questionnaire but with an NT-proBNP level < 125 pg/ml.
Rate of patients with an indeterminate diagnosis of heart failure | 2 months
  Absence of all diagnostic criteria.

SECONDARY OUTCOMES:
Risk factors for heart failure | Day 1
Presence of dyspnea | Day 1
  Evaluation of the main symptoms of heart failure.
Weight gain | Day 1
  Evaluation of the main symptoms of heart failure.
Presence of edema | Day 1
  Evaluation of the main symptoms of heart failure.
Presence of fatigue | Day 1
  Evaluation of the main symptoms of heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel TARTIERE, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (6):
- France (6):
  - Maison de Santé Pluridisciplinaire La Cadière d'Azur, La Cadière-d'Azur, Var
  - Maison de Santé Pluridisciplinaire La Farlède, La Farlède, Var
  - Maison de Santé Pluridisciplinaire Caduceus, La Seyne-sur-Mer, Var
  - Maison de Santé Pluridisciplinaire Beaussetanne, Le Beausset, Var
  - Maison de Santé Pluridisciplinaire Vallée du Gapeau - Sollies-Pont, Solliès-Pont, Var
  - Maison de Santé Pluridisciplinaire Toulon City, Toulon, Var